CLINICAL TRIAL: NCT03546387
Title: Incidence of Neurocognitive Deficits in Patients After Treatment for Retinoblastoma With Multiple Anesthesia Exposures
Brief Title: Determining Whether Multiple Anesthesia Exposures Affect Cognitive Function for Retinoblastoma Patients
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-126
Record Dates: First submitted 2018-05-08; First posted 2018-06-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Retinoblastoma; Retinoblastoma
Keywords: 18-126; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Retinoblastoma | interventions — Wechsler Scales; Memory and Learning Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) — the WISC-V assessment produces a Full Scale IQ (FSIQ) used for primary power consideration in this study. The FSIQ is the most comprehensive global ability score on the WISC-V, and it has been conventionally reported and interpreted as an estimation of overall intellectual ability
Other: California Verbal Learning Test, Children's Version — Used to assess verbal learning and memory in children and adolescents
Other: Beery Developmental Test of Visual Motor Integration, 6th edition — Helps assess visual-motor skills in children and adults.
Other: Grooved Pegboard Test — Measures dexterity
Other: Behavior Assessment System for Children/Parent Report — The Behavior Assessment System for Children/Parent Report is a questionnaire that assesses the social-emotional and behavioral functioning (e.g., anxiety, depression, attention, hyperactivity, adaptability, leadership, social skills, etc.) in children between the ages of 2 and 22 years, and is available in English and Spanish.

SUMMARY:
The purpose of this study is to see if there is a difference between the development of the brain (neurodevelopment) in children who have been treated for retinoblastoma with multiple anesthetic exposures, compared with brain development in children who have never had anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 and < 17 years old

Exclusion Criteria:

* Diagnosis of any secondary disease associated with developmental delay
* History of second cancer diagnosis
* Legal Blindness
* Past surgery of any type, with the exception of enucleation for retinoblastoma
* Past exposure to anesthesia for surgical intervention
* More than one anesthesia encounter for surgical intervention before diagnosis at MSK
* Past External Beam Radiation for treatment of retinoblastoma
* Past systemic chemotherapy
* Non-native speaker of English; however, children whose parents speak only Spanish will be included, because the tests for parents are available in Spanish

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients with retinoblastoma, between 6 and 16 years of age, at MSK.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Comparing scores in neuropsychological testing results | 6 weeks
  The primary outcome is based on the Wechsler Intelligence Scale for Children, 5th edition (WISC-V) measured at follow up. The 5 primary index scores on the WISC-V (Verbal Comprehension, Visual Spatial, Fluid Reasoning, Working Memory, and Processing Speed) are based on 10 subtests and represent intellectual functioning in different cognitive areas. Similar to the FSIQ, the primary index scores are on a standard score metric with a mean of 100 (SD=15). The WISC-V consists of 16 subtests; each subtest is based on a scaled score metric with a mean of 10 and standard deviation (SD) of 3. Performance on these domain-specific subtests will be summarized and analyzed similarly to the FSIQ.

CONTACTS AND LOCATIONS:
Overall Officials: Vittoria Arslan Carlon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org